CLINICAL TRIAL: NCT05750446
Title: Riociguat (BAY 63-2521), a Stimulator of Soluble Guanylate Cyclase (sGC) - Migraine Induction in People With Migraine.
Brief Title: Effect of Riocigaut on Migraine Attack Induction in People With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Messoud Ashina, MD, MD, Ph.D., DMSc., Chief Consultant Neurologist, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H-22041677
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Migraine Without Aura
Keywords: Riociguat; Migraine; Migraine Without Aura; Headache; Pain; Enzyme Activators; Neurologic Manifestations; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Migraine without Aura; Migraine Disorders; Headache; Pain; Neurologic Manifestations | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Riociguat / Placebo (Other): Riociguat or Placebo as oral capsule in randomized order
  Interventions: Drug: Riociguat (BAY 63-2521); Other: Placebo
- Placebo / Riociguat (Other): Riociguat or Placebo as oral capsule in randomized order
  Interventions: Drug: Riociguat (BAY 63-2521); Other: Placebo

INTERVENTIONS:
Drug: Riociguat (BAY 63-2521) — A selective stimulator of soluble guanylate cyclase (sGC)
  Other Names: Adempas
Other: Placebo — Placebo

SUMMARY:
This double-blind, randomized, placebo-controlled cross-over clinical trial aims to investigate the effects of riocigaut on migraine inducing properties in people with migraine.

DETAILED DESCRIPTION:
The investigators believe that activation of sGC could play a role in migraine pathophysiology and propose that stimulation with riociguat causes migraine attacks in people with migraine.

Twenty-one people with migraine are expected to be included. They will participate at a screening visit and, if eligible, on two separate study days, where participants, in a randomized cross-over fashion, will ingest either riociguat (active comparator arm) or placebo (placebo comparator arm), serving as their own controls. On the two separate study days the investigators will measure heart rate, blood pressure and register possible headache/migraine including associated symptoms until 2 hours after intake of riociguat or placebo. At home participants are expected to fill out a headache diary until 12 hours from intake of riociguat or placebo.

ELIGIBILITY:
Inclusion Criteria:

* A history of migraine without aura for ≥ 12 months according to the classification criteria of the International Classification of Headache Disorders 3rd Edition (ICHD-3) criteria.
* An estimated average of between 1-5 migraine attacks per month.
* Ability to provide written informed consent and receive participant privacy and rights information prior to initiation of any study-specific activities.
* Male or female participants aged 18-45 years at screening.
* No migraine preventive treatment at screening or during study conduction.
* Non-smokers

Exclusion Criteria:

* Any current or previous history of other primary or secondary headache disorder(s) apart from tension type headache ≤ 5 days per month.
* Lack of ability to differentiate migraine from other headaches
* Headache within 24 hours before any study related procedures (Provocation Day 1 and Provocation Day 2) - Subjects are however allowed to be re-booked for provocation days according to allowed timelines.
* Any daily medication apart from contraceptives.
* Use of any antihypertensive, nitrates or nitric oxide donors or phosphodiesterase inhibitors, CYP3A4 and P-glycoprotein inhibitors, HIV-proteaseinhibitors, ciclosporin A or CYP1A1-inhibitors, antacida and acid-neutreulizing agents (such as aluminium-/magnesiumhydroxid), CYP3A4-inductors (such as bosentan, phenytoin, carbamazepin, phenobarbital and herbal remedies with perikon).
* Intake of any pro necessitate medication later than 4 times plasma half-life for the specific drug before study start.
* Women of child-bearing potential not currently using safe contraceptives. Women of child-bearing potential does not include hysterectomized women and women who have been in menopause for at least 2 years. Safe contraceptives include either IUD, birth control pills, surgical sterilization of the woman, depositary gestagen, barrier prevention or sexual abstinence.
* Pregnant or breastfeeding women
* Positive pregnancy urine screening on screening day or provocation days.
* A medical history or clinical signs of

  * Hypertension (systolic blood pressure >150mmHg and/or diastolic blood pressure >100mmHg)
  * Hypotension (systolic blood pressure <100mmHg and/or diastolic blood pressure <50mmHg)
* Electrocardiogram (ECG) with any clinically significant abnormalities at screening determined by the investigator, including but not limited to, prolonged PQ or QTc interval, signs of arrythmias, ischemia or left/right ventricle dysfunction/hypertrophy.
* A medical history or clinical signs of pulmo-/cardiovascular disease including cerebrovascular disease.
* A family history of severe cardiac disease.
* A medical history or clinical signs of clinically significant psychiatric illness per investigator opinion.
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior.
* A medical history or clinical signs of substance or alcohol abuse
* A medical history or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the site investigator, would pose a risk to subject safety or interfere with study evaluation, procedures or completion.
* Any history of hypersensitivity to riociguat.
* Subjects who do not want information about crucial pathological findings during the study
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or comply with all required study procedures to the best of the subject and study investigator's knowledge.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Difference in incidence of migraine attacks between riociguat and placebo during a 12-hour observational period after ingestion. | 0-12 hours
  Data will be collected with a questionnaire.

SECONDARY OUTCOMES:
Difference in Area Under the Curve (AUC) values for median headache intensity scores (Numeric Rating Scale (NRS) from 0 to 10, where 0="no pain" versus 1-10="pain") between riociguat and placebo during a 12-hour observational period after ingestion. | 0-12 hours
  Data will be collected with a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Messoud B Ashina, MD, Phd, DMSc, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: No